CLINICAL TRIAL: NCT00952562
Title: The Influence of Vitamin D on Mineral Metabolism, Blood Pressure and Pulse Wave Analysis in Healthy Individuals. A Randomised Double Blinded Placebo Controlled Trial.
Brief Title: The Influence of Vitamin D on Mineral Metabolism, Blood Pressure and Pulse Wave Analysis in Healthy Individuals
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zealand University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 7. juli 2009, version 1
Record Dates: First submitted 2009-08-03; First posted 2009-08-06 (Estimated); Last update posted 2011-08-24 (Estimated); Status verified 2011-08

CONDITIONS: Healthy
Keywords: vitamin d; calcium; blood pressure
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- cholecalciferol (Active Comparator): 3000 IU cholecalciferol per day for 16 weeks
  Interventions: Dietary Supplement: cholecalciferol
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo

INTERVENTIONS:
Dietary Supplement: cholecalciferol — Capsule cholecalciferol 1000 IU, 3 capsules per day for 16 weeks
  Other Names: D3-Vitamin
  Arms: cholecalciferol
Dietary Supplement: placebo — Empty capsules, 3 capsules per day for 16 weeks
  Arms: placebo

SUMMARY:
A randomized placebo controlled trial evaluating the effect of the recently recommended high doses of cholecalciferol (3000 IU/day) on mineral metabolism, blood pressure and pulse wave analysis in healthy individuals.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years old
* p 25OH vitaminD<50nmol/l
* signed informed consent

Exclusion Criteria:

* receiving antihypertensive or antidiabetic treatment
* sarcoidoses
* history of kidney stones
* receiving 1-alfa-hydroxylated vitamin D treatment
* plasma creatinin > 120 micromol/l
* ionised calcium > 1,5 mmol/l
* treatment with calcimimetics
* active malignancy
* intestinal malabsorption
* active pancreatitis
* former hospitalisation due to alcoholic related disease
* using euphoriant drugs
* pregnancy or risk of being pregnant or lactating women
* Known allergy to cholecalciferol capsules

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2009-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

PRIMARY OUTCOMES:
urinary calcium excretion | before and after 16 weeks of intervention

SECONDARY OUTCOMES:
25 hydroxyvitamin D | before and after 16 weeks og treatment
1,25 dihydroxyvitamin D | before and after 16 weeks of treatment
urinary creatinin | before and after 16 weeks of treatment
urinary protein | before and after 16 weeks of treatment
urinary phosphorous | before and after 16 weeks of treatment
p-FGF23 | before and after 16 weeks of treatment
blood pressure | before and after 16 weeks of treatment
pulse wave velocity | before and after 16 weeks of treatment
augmentation index | before and after 16 weeks of treatment
central blood pressure | before and after 16 weeks of treatment
p-phosphate | before and after 16 weeks of treatment
ionised p-calcium | before and after 16 weeks of treatment
p-iPTH | before and after 16 weeks of treatment
alkalic phosphatase | before and after 16 weeks of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Ditte Hansen, MD, Principal Investigator — Zealand University Hospital; Niels Erik Frandsen, MD, Principal Investigator — Zealand University Hospital; Knud Rasmussen, DmSci, Principal Investigator — Zealand University Hospital; Lisbet Brandi, DmSci, Principal Investigator — Zealand University Hospital; Hans Christian Hoeck, DmSci, Principal Investigator — Center for clinical and basic research
Locations (1):
- Roskilde Hospital, Roskilde, Roskilde, Denmark

REFERENCES:
- [Derived] Bressendorff I, Brandi L, Schou M, Nygaard B, Frandsen NE, Rasmussen K, Odum L, Ostergaard OV, Hansen D. The Effect of High Dose Cholecalciferol on Arterial Stiffness and Peripheral and Central Blood Pressure in Healthy Humans: A Randomized Controlled Trial. PLoS One. 2016 Aug 10;11(8):e0160905. doi: 10.1371/journal.pone.0160905. eCollection 2016. PMID 27509187
- [Derived] Nygaard B, Frandsen NE, Brandi L, Rasmussen K, Oestergaard OV, Oedum L, Hoeck HC, Hansen D. Effects of high doses of cholecalciferol in normal subjects: a randomized double-blinded, placebo-controlled trial. PLoS One. 2014 Aug 28;9(8):e102965. doi: 10.1371/journal.pone.0102965. eCollection 2014. PMID 25166750